CLINICAL TRIAL: NCT05904132
Title: Individual Closed-Loop Neuromodulation Therapy for Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joan A Camprodon, MD MPH PhD, Chief, Division of Neuropsychiatry and Neuromodulation, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2023P000785
Record Dates: First submitted 2023-05-22; First posted 2023-06-15 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Healthy Controls (Placebo Comparator)
  Interventions: Device: tACS device
- MCI Subjects (Experimental)
  Interventions: Device: tACS device

INTERVENTIONS:
Device: tACS device — you will receive one of four treatment conditions that include active and sham tACS. The four conditions are the following: (1) closed-loop-tACS (peak-locked), (2) closed-loop-tACS (trough-locked), (3) open-loop tACS, and (4) sham tACS. Although each subject will undergo all four treatments in four separate study visits, the order of the treatments will be randomized

SUMMARY:
The project is a placebo-controlled study that aims to use closed-loop transcranial alternating current stimulation (tACS) to study patients with symptoms of mild cognitive impairment which is likely due to Alzheimer's disease or another form of dementia (AD-MCI). Patients will undergo an EEG and complete some questionnaires and computer tasks during each study visit. The project has the following aims and hypotheses: 1.) To determine the impact of closed-loop 40 Hz tACS on the entrainment of natural gamma rhythms in patients with AD-MCI, 2.) To determine the impact of closed-loop 40 Hz tACS on cognitive performance in patients with AD-MCI, and 3.) To assess the relationship between baseline neurodegenerative burden and impact of tACS. [exploratory]

ELIGIBILITY:
Inclusion Criteria:

* Overall cognitive functional status consistent with amnesic MCI (CDR 0.5) likely due to AD (AD biomarker supported)
* 50-80 years of age
* English native speakers

Exclusion Criteria:

* Known presence of a structural brain lesion (e.g., tumor, cortical infarct)
* Acute or decompensated active medical conditions, including cancer, cardiovascular disease, stroke, congestive heart failure
* Active hematological, renal, pulmonary, endocrine or hepatic disorders
* Longstanding premorbid history (i.e., longer than 10 years) of alcohol or substance abuse with continuous abuse up to and including the time that the symptoms leading to clinical presentation developed
* tACS contraindications (lesions in the scalp, history of seizures)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in the power of entrainment of natural gamma rhythms in patients with AD-MCI. | After a single stimulation session (30 minutes).
  Measured using closed loop 40 Hertz tACS device
Changes in cognitive performance in patients with AD-MCI. | After a single stimulation session (30 minutes).
  Measured using Rey Auditory Verbal Learning Task (RAVLT) which is broken into 6 blocks with each block including a list of 15 words and higher word remembrance in each block indicates a better outcomes, and Face-Name Association Task (FNAT) task where a higher score of matching face to name (out of 60 trials) indicates a better outcome
Changes in gamma power on cognition in patients with AD-MCI including the effect of baseline neurodegenerative burden/biomarkers. [exploratory] | After a single stimulation session (30 minutes).
  Measured using Rey Auditory Verbal Learning Task (RAVLT) which is broken into 6 blocks with each block including a list of 15 words and higher word remembrance in each block indicates a better outcomes, and Face-Name Association Task (FNAT) task where a higher score of matching face to name (out of 60 trials) indicates a better outcome, any MRI/PET scans provided prior to study involvement, and changes in gamma power using closed loop 40 Hertz tACS device

CONTACTS AND LOCATIONS:
Overall Officials: Joan Camprodon, MD, PhD, MPH, Principal Investigator — MGH, Division of Neuropsychiatry and Neuromodulation
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No